CLINICAL TRIAL: NCT04379895
Title: Comparison of Heated vs. Pulsed Radiofrequency Treatment of the Genicular Nerves for Osteoarthritis Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Rimma Geller, MD, Staff pain physician, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0087-19-RMB CTIL
Record Dates: First submitted 2020-03-03; First posted 2020-05-08 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis, Knee
Keywords: treatment; radiofrequency; genicular nerves
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Heated RF ablation (Active Comparator): Patients with OA that will undergo heated RF of the genicular nerves
  Interventions: Device: Radiofrequency ablation
- Pulsed RF ablation (Active Comparator): Patients with OA that will undergo pulsed RF of the genicular nerves
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Radiofrequency ablation — Pulsed or heated RF ablation of the genicular nerves will be done as an Acceptable treatment for OA of the knee

SUMMARY:
This is a prospective, randomised, interventional, double blinded study to compare the clinical outcomes of thermal vs. pulsed radiofrequency (RF) treatment of the genicular nerves in patients with painful osteoarthritis (OA) of the knee.

Population: 60 patients, aged 50 and above, with painful OA of the knee. Interventional measures: Pulsed or heated RF treatment of the genicular nerves of the involved knee.

Outcome measures: primary - fraction of patients experiencing improvement of 50% or higher in their average pain rating during stair climbing.

secondary - improved quality of life

* improved functional capacity
* comparison of side effects and adverse events
* change in the consumption of analgesic medications

DETAILED DESCRIPTION:
Pre-intervention assessment Pain intensity during stairs climbing using VAS 1-100 numerical rating scale. Analgesics consumption. Quality of life using WOMAC questionaires. A physician will further examine them and will enroll them signing an informed concent.

A diagnostic block with lidocaine 2% (2ml for each nerve - total volume of 6ml per knee) of 3 genicular nerves (upper medial and lateral and lower medial branches) will be performed, guided either by ultrasound or by fluoroscopy.

Participants will be asked to fill in a VAS questionnaire shortly (up to one hour) after undergoing the diagnostic blocks.

Participants achieving a relief of >50% in pain intensity during stairs climbing will be considered to have responded to the diagnostic block and will be randomized.

Randomization

Recruited participants will be randomized into two groups:

1. Heated RF ablation
2. Pulsed RF ablation

Blinding Both the patient and the assessing physician will be blinded to the group to which the patient has been allocated. The physicians performing the treatment will be blinded as well.

Intervention

Heated RF ablation of the genicular nerves will be performed as follows:

1. In the supine position, aseptic preparation of the skin and sterile coverage of the procedure area will take place.
2. After the administration of local anesthesia to the skin with lidocain 2% (1-1.5cc for each injection site, fluoroscopy guided placement of three 22 gauge 50mm or 100mm straight RF cannulas in the proximity of 3 of the genicular nerves: 2 on both sides of the distal femoral shaft-epiphysis border and one on the medial proximal tibial epiphyseal-shaft border.
3. Sensory stimulation at 50 Hertz will be used to test the proper position of the needle, expected to generate paresthesia in the distribution of the affected nerve, at a voltage in the range of 0.3-0.8 Volts. Motor stimulation at 2 Hz will be used to exclude proximity of the cannula to motor nerves.
4. 1 ml of 2% lidocaine will be injected into each cannula.
5. 180 sec 80 degrees heated RF ablation of the nerves will be performed. Needles will be left in place for additional 420 seconds to match the treatment duration of the pulsed RF group.
6. Injection of a total amount of 80 mg methylprednisolone and lidocaine 2% 2cc to the 3 intervention sites.

Pulsed RF ablation of the genicular nerves will be performed similarly to the heated RF ablation with the only difference being that the treatment will include a 600 sec of 42 degrees heating of the three-genicular nerves.

Blinding Both the patient the assessing and performing physicians will be blinded to the group to which the patient has been allocated.

Post-procedural assessment Participants will be assessed 3 days and 30 days after the procedure (phone questionnaires) and a clinical follow-up visits in 3 and 6 months after the procedure.

The assessment will include:

1. Two telephone interviews, in which the patient will report the average severity of pain on a 1 to 100 numerical rating scale and will fill up a WOMAC questionnaire regarding the treated knee in the prior 24 hours.
2. Two clinic follow-up visit, during which the patients will fill-in a questionnaire of pain intensity after stairs climbing using VAS 1-100 numerical rating, analgesic consumption, quality of life measures using the WOMAC questionaire. Questionnaires filling-in will be aided and supervised by research assistants blinded to the intervention the participants have received.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically proven OA of knee with a 2. Kellgren-Lawrence scale (K-L score) of 3 to 4.
* Clinically proven OA of knee with an Oxford knee score of 0 to 30 (representing moderate to severe OA).
* Chronic knee pain due to the OA of knee (>3 months) of at least moderate severity by a Visual Analogue Scale (VAS) 4 and above.
* Signed informed consent

Exclusion Criteria:

* Acute knee pain
* Disease that preclude per clinician decision interventional treatment.
* Allergic reaction to the injected substances (triamcinolone, lidocaine)
* Injections to the knee during the 3 months preceding recruitment
* Distorted knee intervention due to any cause, which interferes with the radiological identification of targeted RF sites.
* Anticoagulation treatment that cannot be stopped.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Knee pain reduction | 3 months
  Reduction in knee pain during stairs climbing by at least 50% in a 1-10 Numerical Rating Scale (NRS) pain severity score and a comparison between the 2 techniques outcomes.

SECONDARY OUTCOMES:
quality of life measurements improvement | 3 months
  Improvement in quality of life measures using The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questionaires
Adverse events | 3 months
  Comparison of the two groups

REFERENCES:
- [Background] Gupta A, Huettner DP, Dukewich M. Comparative Effectiveness Review of Cooled Versus Pulsed Radiofrequency Ablation for the Treatment of Knee Osteoarthritis: A Systematic Review. Pain Physician. 2017 Mar;20(3):155-171. PMID 28339430
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] Cohen SP, Peterlin BL, Fulton L, Neely ET, Kurihara C, Gupta A, Mali J, Fu DC, Jacobs MB, Plunkett AR, Verdun AJ, Stojanovic MP, Hanling S, Constantinescu O, White RL, McLean BC, Pasquina PF, Zhao Z. Randomized, double-blind, comparative-effectiveness study comparing pulsed radiofrequency to steroid injections for occipital neuralgia or migraine with occipital nerve tenderness. Pain. 2015 Dec;156(12):2585-2594. doi: 10.1097/j.pain.0000000000000373. PMID 26447705
- [Background] Kroll HR, Kim D, Danic MJ, Sankey SS, Gariwala M, Brown M. A randomized, double-blind, prospective study comparing the efficacy of continuous versus pulsed radiofrequency in the treatment of lumbar facet syndrome. J Clin Anesth. 2008 Nov;20(7):534-7. doi: 10.1016/j.jclinane.2008.05.021. PMID 19041042
- [Background] Protzman NM, Gyi J, Malhotra AD, Kooch JE. Examining the feasibility of radiofrequency treatment for chronic knee pain after total knee arthroplasty. PM R. 2014 Apr;6(4):373-6. doi: 10.1016/j.pmrj.2013.10.003. Epub 2013 Dec 27. PMID 24373908
- [Background] Iannaccone F, Dixon S, Kaufman A. A Review of Long-Term Pain Relief after Genicular Nerve Radiofrequency Ablation in Chronic Knee Osteoarthritis. Pain Physician. 2017 Mar;20(3):E437-E444. PMID 28339444